CLINICAL TRIAL: NCT00941707
Title: A Phase IIa Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of JNJ-38518168 in Patients With Active Rheumatoid Arthritis Despite Methotrexate Therapy With Synovial Biopsy Substudy
Brief Title: An Efficacy and Safety Study of JNJ-38518168 in Adult Participants With Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to a single, unexpected serious event, the trial was stopped.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016414; 2009-012118-27 (EudraCT Number); 38518168ARA2001
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; JNJ-38518168
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JNJ-38518168 (Experimental)
  Interventions: Drug: JNJ 38518168
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ 38518168 — JNJ-38518168 100 milligram (mg) capsules orally (by mouth) once daily for 12 weeks.
  Arms: JNJ-38518168
Drug: Placebo — Placebo capsules matching to JNJ-38518168 orally once daily for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, tolerability and safety of JNJ-38518168 compared with placebo in adult participants with active rheumatoid arthritis (long time systemic disease of the joints, marked by inflammatory changes in the synovial membranes and bones) despite methotrexate (MTX) therapy.

DETAILED DESCRIPTION:
This is a multi-center (when more than 1 hospital or medical school team work on a medical research study), randomized (the study drug is assigned by chance), double-blind (neither physician nor participant knows the treatment that the participant receives), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect) and parallel-group (each group of participants will be treated at the same time) study. The study will consist of 3 phases; Screening phase (3 weeks), Treatment phase (12 weeks) and Follow-up phase (4 weeks). Each participant will be enrolled in the study for approximately 19 weeks. Participants with active rheumatoid arthritis despite MTX therapy will receive JNJ-38518168, 100 milligram (mg) per day or matching placebo capsules once daily for 12 weeks. Efficacy will be primarily evaluated by change from Baseline in disease activity index score C-reactive protein at Week 12. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with rheumatoid arthritis (RA) according to the revised 1987 criteria of the ARA (Arnett et al, 1988) for at least 6 months at Screening
* Participants who have been treated with and tolerated methotrexate (MTX) treatment at dosages from 7.5 to 25 milligram (mg) per week inclusive, for a minimum of 4 months before Screening
* Participants if using non-steroidal anti-inflammatory drugs (NSAIDs) or other analgesics (drug used to control pain) regularly for RA, participants must have been on a stable dose for at least 2 weeks before the first dose of study medication
* Participants if using oral corticosteroids (compounds, usually hormonal, taken orally [by mouth] in order to block ovulation [discharge of an egg from the ovary] and prevent the occurrence of pregnancy [carrying an unborn baby]), must be on a stable dose of less than or equal to 10 mg per day of prednisone or another oral corticosteroid for at least 4 weeks before the first dose of study medication and continue with the same dose throughout the study. If not using corticosteroids at study initiation, the participant must have not received any oral corticosteroids for at least 4 weeks before the first dose of study medication
* Participants currently treated with folic acid at a minimum dose of 5 mg per week

Exclusion Criteria:

* Participants having inflammatory disease other than RA
* Participant who have used any of the following medications: D-penicillamine, hydroxychloroquine, chloroquine, oral or parenteral gold salts, sulfasalazine, leflunomide, azathioprine, cyclosporine, tacrolimus, and mycophenolatemofetil
* Participant who have received intra-articular, intramuscular (into the muscle), or intravenous (into the vein) corticosteroids, including adrenocorticotropic hormone (hormone made by the brain that activates the adrenal glands) within 4 weeks before the first dose of the study medication
* Participants who have been treated with any other investigational drug or medical device within 4 weeks or 5 half-lives of the drug, whichever is longer before the first dose of study medication
* Participants who have undergone surgical treatments for RA including synoviectomy (surgical removal of a part of the synovial membrane of a joint) and arthroplasty (surgery to fix a joint) within 3 months before the first dose of study medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Disease Activity Index Score (DAS28) C-Reactive Protein (CRP) at Week 12 | Baseline and Week 12
  The DAS28 based on CRP is a statistically derived index combining tender joints (28 joints), swollen joints (28 joints), CRP and participant's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst.

SECONDARY OUTCOMES:
Percentage of Participants With DAS28 (CRP) Response | Week 12
  The DAS28 based on CRP is a statistically derived index combining tender joints (28 joints), swollen joints (28 joints), CRP and participant's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, MCP1 to MCP5, proximal PIP, PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst.
Percentage of Participants With DAS28 (ESR) Response | Week 12
  The DAS28 based on erythrocyte sedimentation rate (ESR) is a statistically derived index combining tender joints (28 joints), swollen joints (28 joints), ESR and global health (GH). The DAS28-ESR is expressed on a score on a scale with the minimum score=0 (best) to maximum score=10 (worst).
Change From Baseline in DAS28 (ESR) Score at Week 12 | Baseline and Week 12
  The DAS28 based on ESR is a statistically derived index combining tender joints (28 joints), swollen joints (28 joints), ESR, and GH. The DAS28-ESR is expressed on a score on a scale with the minimum score=0 (best) to maximum score=10 (worst).
Percentage of Participants Achieving American College of Rheumatology (ACR20) Response | Week 12
  The ACR20 response is defined as more than or equal to (>=) 20 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=20 percent improvement in 3 of following 5 assessments: participant's assessment of pain using Visual Analog Scale (VAS; 0-10 millimeter (mm), 0 mm=no pain and 10 mm=worst possible pain), participant's global assessment of disease activity by using VAS, physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI) and CRP.
Percentage of Participants Achieving ACR50 Response | Week 12
  The ACR50 response is defined as >=0 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=50 percent improvement in 3 of the following 5 assessments: participant's assessment of pain using VAS, participant's global assessment of disease activity by using VAS, physician's global assessment of disease activity using VAS, participant's assessment of physical function as measured by HAQ-DI and CRP.
ACR-N Index Score | Week 12
  The ACR-N Index of improvement is defined as the minimum of the following 3 criteria: percent improvement from Baseline in tender joint counts, percent improvement from Baseline in swollen joint counts and median percent improvement from Baseline for the following 5 assessments: participant's assessment of pain using VAS, participant's global assessment of disease activity using VAS, physician's global assessment of disease activity using VAS, participant's assessment of physical function as measured by HAQ-DI and CRP. Negative numbers indicate worsening.
Change From Baseline in HAQ-DI at Week 12 | Baseline and Week 12
  The HAQ-DI is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping and activities of daily living). Responses in each functional area are scored from 0 to 3 (0=no difficulty and 3=inability to perform a task in that area).
Change From Baseline in Participant's Assessment of Pain at Week 12 | Baseline and Week 12
  Participants will assess their average pain on a VAS. The scale ranges from 0 mm to 100 mm, (0 mm=no pain to 100 mm=worst possible pain).
Change From Baseline in Physician's Global Assessment of Disease Activity at Week 12 | Baseline and Week 12
  The Investigator's global disease assessments will be recorded on a VAS. The scale for the Investigator's assessments ranges from 0 mm to 100 mm (0 mm=no arthritis activity, 100 mm=extremely active arthritis).
Change From Baseline in Patient's Global Assessment of Disease Activity at Week 12 | Baseline and Week 12
  The participant's global disease assessments will be recorded on a VAS. The scale ranges from 0 mm to 100 mm (0 mm=very well to 100 mm=very poor).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (34):
- Liège, Belgium
- Czechia (5):
  - Brno
  - Kladno
  - Prague
  - Uherské Hradiště
  - Zlín
- Dublin, Ireland
- Amsterdam-Zuidoost, Netherlands
- Poland (5):
  - Bialystok
  - Bydgoszcz
  - Elblag
  - Lublin
  - Torun
- Russia (7):
  - Kemerovo
  - Moscow
  - Novosibirsk
  - Petrozavodsk
  - Saint Petersburg
  - Yaroslavl
  - Yekaterinburg
- South Korea (3):
  - Pucheon
  - Seoul
  - Suwon
- Spain (4):
  - Barcelona
  - Guadalajara
  - Santiago de Compostela
  - Seville
- Taiwan (3):
  - Changhua
  - Taichung
  - Taipei
- United Kingdom (4):
  - London
  - Middlesbrough
  - Salford
  - Wigan